CLINICAL TRIAL: NCT01995643
Title: Effect of Grape Seed Extract on Modulation of Oxidative Stress/ Inflammation/ Insulin Sensitivity Induced by High Fat-carbohydrate Meal in Healthy Human Subjects
Brief Title: Acute Effects of Grape Seed Extract on Insulin Sensitivity and Oxidative Stress and Inflammation Markers.
Acronym: GSE2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 2013-114
Record Dates: First submitted 2013-11-21; First posted 2013-11-26 (Estimated); Last update posted 2021-07-27 (Actual); Status verified 2020-07

CONDITIONS: Polyphenolic Compounds and Metabolism
Keywords: Grape seed extract; Polyphenols; Insulin; Oxidative stress Marker; Inflammatory marker; Healthy human
MeSH Terms: conditions — Insulin Resistance | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Capsule (Active Comparator): Grape Seed Extract Capsule: 300 mg
  Interventions: Dietary Supplement: Active Capsule
- Placebo Capsule (Placebo Comparator): Placebo Capsule: Maltodextrin
  Interventions: Dietary Supplement: Placebo Capsule

INTERVENTIONS:
Dietary Supplement: Active Capsule — GSE Capsule
  Arms: Active Capsule
Dietary Supplement: Placebo Capsule — Placebo Capsule
  Arms: Placebo Capsule

SUMMARY:
The proposed study aims to investigate that consumption of grape seed extract (GSE) would improve antioxidant status and impaired insulin action following consumption of a pro-oxidative high carbohydrate, high fat (HCHF) meal in healthy human subjects.

DETAILED DESCRIPTION:
This study is a single-center, double blind, placebo-controlled, randomized, 2-arm, 2-sequence, crossover study

A planned sample size of 15 will be recruited into the study. This study will require one initial screening, one pre-study visit, two 6-hour study visits. The study will take 2-5 weeks per subject to complete.

The initial screening visit will provide subjects an Institutional Review Board approved consent document and determine subject eligibility through BMI calculated from height and weight measurements, vital signs, fasting blood glucose test (finger prick), lipid profiles (3 ml blood sampling via a butterfly needle device) and completion of a questionnaire related to general eating, health, and exercise habits.

If subjects are willing and eligible to participate, a 3-day food record (2 weekdays and 1 weekend day) will be instructed at the initial screening visit and collected at the pre-study visit to assess subjects' usual dietary intake pattern. After reviewing food records, subjects will be instructed to avoid any grapes, grape products, berries, berry products throughout the study and strictly follow a limited polyphenolic diet for 3 days prior to each 6-hr study visit, while maintaining their usual diet pattern and physical activity. Prior to each study visit, subject will be advised to have the same or similar dinner meal to control the second meal effect from food and beverage intake of the night before each study visit.

Subjects will arrive at the center after ~10 hours overnight fasting, well hydrated and rested. Each study visit will require blood draws throughout the visit. After pre-study procedures (height, weight, waist circumferences, vital sign, and fasting blood glucose test), a registered nurse will place a catheter in subject's arm for the purpose of multiple blood sample collections and collect fasting blood sample. During each study visit, subject will take one of the two capsules right after fasting blood draw), based on randomization sequences (either 1 grape seed extract capsule or 1 placebo capsule). One hour after administration of the assigned capsule, blood samples will be collected. And a standard high carbohydrate and high fat breakfast meal will be served and subject will have blood draws at designated time up to 5 hours.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 20 to 65 years old
* Body Mass Index (BMI) range from 18.5 to 24.9 kg/m2; exception BMI 18.5 to 23 kg/m2 for Asian population
* Fasting blood glucose concentration < 110 mg/dL
* Fasting LDL-cholesterol <180 mg/dL
* Fasting Total cholesterol and Fasting Triglycerides < 250 mg/dL
* Weight stable: not gained or lost weight +/- 5 lbs in previous 3 months
* Non-smokers
* No clinical evidence of cardiovascular, metabolic, respiratory, renal, gastrointestinal or hepatic disease
* Not taking any medications or dietary supplements that would interfere with outcomes of the study, i.e. lipid lowering medications, anti-inflammatory drugs, fish oil, probiotics, grape seed supplement, etc…If anti-inflammation and/or antibiotic medications/supplements are taken, subjects may qualify if go off these medications/supplements 30 days wash-out before entering the study.
* Able to provide informed consent
* Able to comply and perform the procedures requested by the protocol

Exclusion Criteria:

* Past smokers: abstinence for less than 2 years
* Men and women who smoke
* Men and women with known or suspected food intolerance, allergies or hypersensitivity to the study materials or closely related compound or any their stated ingredients.
* Men and women known to have/diagnosed with diabetes mellitus
* Men and women who have fasting blood glucose concentrations ≥110 mg/dL
* Men and women who have uncontrolled blood pressure >140 mmHg/90 mmHg
* Men and women with documented vascular disease, e.g., heart failure, myocardial infarction, stroke, angina, related surgeries.
* Men and women with cancer other than non-melanoma skin cancer in previous 5 years.
* Men and women who are taking medication or dietary supplements that may interfere with the outcomes of the study; e.g., antioxidant supplements, anti-inflammation, lipid lowering medication. Subjects may choose to go off dietary supplements (requires 30 days washout).
* Men and women who are taking blood pressure lowering medication that may interfere the outcomes of the study; e.g. diuretics.
* Men and women who have donated blood within 3 months of the screening visit and blood donors/participants for whom participation in this study will result in having donated more than 1500 milliliters of blood in the previous 12 months.
* Men and women who are vegetarians or vegans
* Substance (alcohol or drug) abuse within the last 2 years.
* Excessive coffee and tea consumers (> 4 cups/day)
* Men and women who do excessive exercise regularly or athlete
* Unstable weight: gained or lost weight +/- 5 lbs in previous 3 months
* Women who are known to be pregnant or who are intending to become pregnant over the course of the study
* Women who are lactating

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2014-08-01 (Actual); Study Completion 2014-08-30 (Actual)

PRIMARY OUTCOMES:
Changes in insulin and glucose concentrations over 6 hours after the Grape Seed Extract Capsule administration | 6 hours
  The timing influence of the Grape Seed Extract administration on insulin and glucose concentrations in relative to the standard meal intake (1 hour before the meal and 5 hours after the meal)

SECONDARY OUTCOMES:
Changes in oxidative stress markers and inflammatory markers over 6 hours after the Grape Seed Extract Capsule administration | 6 hours
  The timing influence of grape seed extract administration on oxidative stress markers and inflammatory markers in relative to the standard meal intake (1 hour before the meal and 5 hours after the meal)

CONTACTS AND LOCATIONS:
Overall Officials: Indika Edirisinghe, Ph.D, Principal Investigator — Institute for Food Safety and Health; Britt Burton-Freeman, Ph.D, MS, Study Chair — Institute for Food Safety and Health
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States